CLINICAL TRIAL: NCT01558076
Title: Longitudinal Changes in Exercise Capacity in Children and Young Adults With Sickle Cell Anemia
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert I. Liem, Professor of Pediatrics, Attending Physician - Hematology-Oncology, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2011-14565; 1K23HL094376 (NIH)
Record Dates: First submitted 2012-03-13; First posted 2012-03-20 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle cell anemia; exercise testing; cardiopulmonary disease
MeSH Terms: conditions — Anemia, Sickle Cell; Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects with sickle cell anemia: 60 subjects with sickle cell anemia will be enrolled on the study.
- 30 healthy controls: 30 controls without sickle cell anemia or sickle cell trait will be enrolled on the study.

SUMMARY:
The purpose of this study is to use comprehensive exercise testing to examine longitudinal changes in exercise capacity over a 2 year period in children and young adults with sickle cell anemia.

DETAILED DESCRIPTION:
Although the burden of sickle cell anemia (SCA) on affected individuals is significant, few studies have examined the influence of having SCA on such measures of physical function as exercise capacity. Moreover, the physiologic basis of poor physical functioning in children with SCA is unknown and has not been studied extensively. The purpose of this proposal is to use cardiopulmonary exercise testing (CPET) to gain a comprehensive understanding of longitudinal changes in exercise capacity, and the effect of poor exercise capacity on quality of life in children and young adults with SCA. The specific aims of this project are to: 1) Measure peak oxygen consumption (VO2), the reference standard for exercise capacity, in children and young adults with SCA classified by primary pathophysiologic contributor to their decreased exercise capacity, and 2) compare results of this exercise test with the results of previously completed exercise tests to determine longitudinal changes in exercise capacity. These aims will be performed in 60 subjects with SCA and 30 matched controls who participated in a previous study, IRB# 2009-13659; "The Physiologic Assessment of Exercise Capacity in Pediatric Sickle Cell Anemia". In a secondary analysis, we will also study the participants quality of life using a set of validated questionnaires. This study is essential because it will address several areas of exercise capacity, including the longterm effects of physiologic contributors to exercise limitation, that remain fundamental knowledge gaps in SCA.

ELIGIBILITY:
Inclusion Criteria:

1. age 8 to 21 years old; AND
2. Hb SS or S-β0 thalassemia disease, confirmed by hemoglobin analysis; AND
3. Previously participated in ClinicalTrials.gov ID: NCT01527799

Exclusion Criteria:

1. inability to perform maximal testing due to physical limitation (e.g. stroke or avascular necrosis); OR
2. history of exercise-induced syncope or arrhythmias. Subjects will wait at least 2 weeks following any vaso-occlusive pain episode and 12 weeks following any disease-related complication requiring transfusion support. Individuals on hydroxyurea will be eligible. A total of 30 controls without SCA or sickle cell trait will be matched for age, sex and race and recruited from the siblings, friends or relatives of subjects enrolled on this study

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sickle cell anemia patients followed at Children's Memorial Hospital. Healthy controls without sickle cell anemia or sickle cell trait are recruited through flyers posted in Children's Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
VO2 max on cardiopulmonary exercise test | Baseline

SECONDARY OUTCOMES:
Quality of life questionnaires | Baseline
Echocardiogram | Baseline
Dual Energy X-ray Absorbtiometry | Baseline
Pulmonary Function Test | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert I Liem, MD MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States